CLINICAL TRIAL: NCT06649201
Title: Vulvovaginal Graft-versus-Host Disease: Diagnosis and Microbiome Evaluation
Status: Recruiting | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CASE2Z24
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Graft Vs Host Disease; Vulvovaginal Signs and Symptoms
Keywords: Allogeneic Hematopoietic Cell Transplantation; Vaginal Microbiome; GVHD; HCT; Vulvovaginal GVHD; Vulvovaginal graft-versus-host disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microbiome samples will be collected by a provider and will be transported to the Genomic Medicine Biorepository Core laboratory. All samples will be de-identified, coded and stored in the Genomic Medicine Biorepository indefinitely using established practice of the Genomic Medicine Biorepository Core. Additional samples for gonorrhea, chlamydia, bacterial vaginosis, candidiasis and trichomoniasis will be transported to the general Cleveland Clinic Laboratory and processed there using their standard protocols per clinic standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic HCT participants: The cohort will be comprised of participants undergoing allogeneic HCT at the Cleveland Clinic.
  Interventions: Other: Vulvovaginal Symptom Questionnaire; Diagnostic Test: Vaginal Microbiome Evaluation

INTERVENTIONS:
Other: Vulvovaginal Symptom Questionnaire — Participants will undergo assessment of vulvovaginal symptoms via the vulvovaginal questionnaire once pre-transplant, six months, and develop months post-transplant.
Diagnostic Test: Vaginal Microbiome Evaluation — A vaginal microbiome evaluation will be performed via vaginal exam by a gynecologist with collection of vaginal samples once pre-transplant, six months, and twelve months post-transplant.

SUMMARY:
The goal of this observational study is to investigate the development of vulvovaginal graft-versus-host- disease (GVHD), an under-reported and under-recognized manifestation of chronic GVHD. This study aims to characterize the vaginal microbiome in participants undergoing allogeneic hematopoietic cell transplantation (HCT). The main questions it aims to answer are:

* Is the vaginal microbiome altered during allogeneic HCT?
* What changes may help researchers understand the development of vulvovaginal GVHD?

Participants will be asked to undergo an assessment of vulvovaginal symptoms through a vulvovaginal symptom questionnaire once pre-transplant, 6 months post-transplant, and twelve12 months post- transplant. Participants will also be asked to undergo a vaginal microbiome (collection of bacteria, fungi, and viruses that live on our bodies) evaluation through a vaginal exam performed by a gynecologist with collection of vaginal samples once pre-transplant and again six months post-treatment and twelve months post-transplant. If a participant develops symptoms of vulvovaginal GVHD at any point in time during the post-transplant follow up, the participant may partake in additional vaginal exams to diagnose GVHD at the time of symptom onset.

DETAILED DESCRIPTION:
Recent advances in technologies including high throughput metagenomic 16S rRNA gene sequencing have revealed a larger, more complex picture of the bacterial diversity in the genital tract and unique microbial communities not previously recognized among the known vaginal flora categories. Little is known about how the vaginal microbiome protects the female genital tract or other roles it may have, including interacting with the microbiota of other body sites and subsequent inflammatory responses. Alteration of vaginal flora may play a part in the pathogenesis of diseases by modulating immunity or increasing the growth of pathogenic strains. Recent research has been conducted regarding changes in the vaginal microbiome during various infectious and inflammatory states such as bacterial vaginosis, pelvic inflammatory disease, sexually transmitted infectious, and pregnancy. However, the vaginal microbiome during allogeneic HCT and development of genital GVHD has yet to be examined. Thus, the role of the vaginal microbiome in the development of genital GVHD is a critical area of study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants planning to undergo allogeneic HCT for any disease indication, OR, female participants who have already received HCT and have developed vulvovaginal GVHD during their post-transplant follow-up period
* All conditioning regimens (myeloablative or reduced intensity) will be included.
* All donor sources (HLA matched/mismatched related, unrelated, umbilical cord, haploidentical) will be included.
* All graft sources (bone marrow or peripheral blood stem cells) will be included.
* All GVHD prophylaxis regimens will be included.
* Aged 18-70.
* English speaking and able to sign written informed consent.
* Participants agree to a vaginal gynecologic exam.
* Co-enrollment on other clinical trials will be allowed.

Exclusion Criteria:

* Participants who decline or unable to undergo vaginal gynecologic exam due to any discomfort or pain.
* Any concurrent medical, psychiatric or other illness in which the provider believes the participants may not be able to comply with study assessments.
* Participants with a current diagnosis of a sexually transmitted infection (STI) (Herpes Simplex Virus, Gonorrhea, Chlamydia, Trichomonas,) or a history of previously untreated STI which may incite inflammation that will impact the microbiome.
* Participants with a history of lichen sclerosis, lichen planus, pre-transplant.
* Participants with a history or current diagnosis of vaginal or vulvar malignancy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female participants undergoing allogenic HCT will be recruited from the Blood and Marrow Transplant Program at the Cleveland Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Characterize the vaginal microbiome profile of female participants undergoing allogeneic HCT | Up to twelve months post-transplant
  A primary objective of this study is to characterize the vaginal microbiome and in female participants undergoing allogeneic HCT.
Characterize the change in vaginal microbiome profile of female participants undergoing allogeneic HCT | Up to twelve months post-transplant
  A primary objective of this study is to characterize the vaginal microbiome change in female participants undergoing allogeneic HCT.
Incidence of vulvovaginal GVHD | Up to twelve months post-transplant
  A primary objective is to measure the incidence of vulvovaginal GVHD in this cohort.

SECONDARY OUTCOMES:
Characterize the differences in vaginal microbiome between participants who develop vulvovaginal GVHS versus those who do not | Up to twelve months post-transplant
  The secondary objective is to investigate differences in vaginal microbiome between participants who develop vulvovaginal GVHD and those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Betty K Hamilton, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No